CLINICAL TRIAL: NCT02523859
Title: A Randomized, Single-blind, Propofol-controlled Phase III Study Evaluating the Efficacy and Safety of Remimazolam in GA in Adult Patients Undergoing Cardiac Surgery, Including Follow-up Sedation in the Post-anesthesia Care Unit/ICU
Brief Title: Study of the Efficacy and Safety of Remimazolam in General Anesthesia in Adults Undergoing Cardiac Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Paion UK Ltd. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNS7056-011
Record Dates: First submitted 2015-08-11; First posted 2015-08-14 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Propofol; remimazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Propofol for induction will be given as a bolus administered manually at 2.0-2.5 mg/kg slowly over approximately 1 minute. Immediately after the propofol bolus for induction has been given, propofol maintenance will be started at a dose of 3.0-9.0 mg/kg/hr and adjusted as needed.
  Interventions: Drug: Propofol
- Remimazolam (Experimental): Remimazolam for induction will be given at 6.0 mg/kg/hr, which can be increased to 12.0 mg/kg/hr for one minute if loss of consciousness is not reached after 3 minutes. Immediately after the remimazolam dose for induction has been given, remimazolam maintenance will be given at 1.0 mg/kg/hr and adjusted by down-titration or up-titration to a maximum of 3.0 mg/kg/hr.
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Propofol — Hypnotic drug used for anesthesia
  Other Names: Diprivan
  Arms: Propofol
Drug: Remimazolam — Benzodiazepine being developed for sedation and anesthesia.
  Other Names: CNS7056
  Arms: Remimazolam

SUMMARY:
This study investigates the use of remimazolam as a sedative/hypnotic in general anesthesia. Remimazolam or propofol will be administered together with fentanyl/sufentanil/remifentanil as opioid analgesics and a neuromuscular blocker.

In total, 530 patients will be randomized. This group of 530 patients will be split randomly into 2 groups as follows:

• 106 patients will be randomized to induction with propofol plus fentanyl or sufentanil or remifentanil and a neuromuscular blocker. Throughout maintenance, the patients will receive propofol and remifentanil until weaning from the mechanical ventilation on the ICU or PACU within 24 hours after induction.

Afterwards, sedation with propofol as study medication has to be ended. If necessary, the sedation is to be continued with the hospital's own supplies (propofol or other sedative).

• 424 patients will be randomized to induction with remimazolam 6.0 mg/kg/hr together with fentanyl or sufentanil or remifentanil and a neuromuscular blocker. Throughout maintenance, the patients will receive remimazolam and remifentanil until weaning from the mechanical ventilation on the ICU or PACU within 24 hours after induction.

The primary endpoint is successful sedation is defined as a Narcotrend index of 60 or less during at least 85% of the maintenance time and no rescue sedative medication administered. The maintenance starts at arrival at the operation theater and ends with the completion of the last skin suture.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for major non-emergency cardiac surgery, i.e. surgery assumed to require more than 2 hours of maintenance of general anesthesia and to require the use of extracorporeal circulation, including coronary bypass(es), valve replacement(s), and associated procedures and on-pump minimal invasive surgery
2. Scheduled to receive mechanical ventilation via tracheal intubation (oropharyngeal or nasotracheal)
3. Age at least 18 years
4. Body mass index 18 to ≤40 kg/m2
5. Willingness and ability to give informed consent, to understand, participate and comply with all study requirements
6. For women of childbearing potential: negative pregnancy test (serum or urine strip) as well as using a highly effective method of birth control. Such methods include:
7. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, with the following routes of administration: oral, intravaginal, transdermal
8. Progestogen-only hormonal contraception associated with inhibition of ovulation, with the following routes of administration: oral, injectable, implantable
9. Intrauterine device
10. Intrauterine hormone-releasing system
11. Bilateral tubal occlusion
12. Sexual abstinence A woman was considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods included hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

Exclusion Criteria:

1. Re-do cardiac surgery
2. Surgical procedures that comprised the use of drugs and/or devices that were not approved for marketing
3. Severe tricuspidal insufficiency (III grade)
4. Planned cooling of the patient's body below 32ºC
5. History of or planned stop of circulation, e.g. due to repair of type A dissection of aorta or removal of thrombi from pulmonary artery
6. Planned to receive epidural/spinal anesthesia together with general anesthesia
7. Evidence of uncontrolled hepatic, central nervous system, respiratory, or metabolic dysfunction, or other clinically significant findings at screening that, in the investigator's or medical monitor's opinion, excluded patients from the study
8. Poorly controlled hypertension (e.g. systolic blood pressure ≥160 mmHg under antihypertensive medication at screening)
9. Patients with severe renal insufficiency or end-stage renal disease (creatinine clearance below 30 mL/min or estimated glomerular filtration rate below 30 mL/min/1.73 m2). Measuring only one of both parameters was sufficient to assess the eligibility of a patient.
10. Patients with clinically uncontrolled coagulation abnormalities, or with coagulation abnormalities not under adequate treatment
11. Patients scheduled for heart or lung transplantation
12. Patients with infectious cardiac disorders (e.g. endocarditis, myocarditis)
13. Patients with sepsis
14. Emergency surgery, status of shock or coma
15. Patients with an ejection fraction from the left ventricle of less than 20%
16. Patients with acute right heart failure
17. Pre-operative use of phosphodiesterase 3 inhibitors
18. Patients with a history of resuscitation
19. Known resistance to benzodiazepines or history of paradoxical effects after administration of benzodiazepines
20. History of hypersensitivity to benzodiazepines, propofol, remifentanil hydrochloride, neuromuscular blockers, flumazenil or other anesthetic agents
21. Use of benzodiazepines within 5 times their half-life or 5 times the half-life of their active metabolites. Exception: Pre-medication with a benzodiazepine according to local standards was allowed.
22. Epilepsy
23. Myasthenia gravis or myasthenic syndrome
24. History of any severe allergy defined as urticaria, angioedema or anaphylaxis
25. Dependence from drugs or history of drug abuse
26. Dependence from alcohol or history of alcohol abuse within the last 5 years
27. Acute alcoholic intoxication or ethanol intake within 48 hours prior to surgery
28. Acute narrow-angle glaucoma
29. Female patients of childbearing potential without acceptable method of birth control (for definitions: see inclusion criterion 6).
30. Pregnant or breast-feeding female patients
31. Patients in receipt of any investigational drug within 30 days or less than 7 half-lives (whichever was longer) before the start of the study, or scheduled to receive one during the study period.
32. Administration of remimazolam in the past
33. Patients unable to communicate with the investigator as required for the study
34. Other reasons that, according to the investigator, excluded the patient from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Success of Procedure | During maintenance phase of operation - between arrival at operation theatre and completion of last skin suture (estimated up to 24 hours).
  A narcotrend index of 60 or less during at least 85% of the maintenance time and no rescue sedative medication administered.

SECONDARY OUTCOMES:
Hemodynamic stability | From the start of study medication until completion of the last skin suture (estimated up to 24 hours).
  Expressed as the amount of norepinephrine used.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Probst, MD, Principal Investigator — Herzzentrum Leipzig GmbH
Locations (1):
- Herzzentrum Leipzig GmbH, Leipzig, Germany